CLINICAL TRIAL: NCT01006642
Title: Minimal Changes of Gastric Mucosal Barrier in the Pathophysiologic Mechanisms of Functional Dyspepsia
Brief Title: Mucosal Barrier Defects in Functional Dyspepsia by Confocal Laser Endomicroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Yan-Qing Li, Department of Gastroenterology, Qilu Hospital, Shandong University
Other Study IDs: 2009SDU-QILU-G04
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies during endoscopy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy controls: Asymptomatic individuals admitted for health surveillance or patients for follow up after polypectomy.
- Functional dyspepsia-EPS: Functional dyspepsia-EPS(epigastric pain syndrome) Patients admitted to outpatient department with symptoms meeting ROME III criteria
- Functional dyspepsia-PDS: Functional dyspepsia-PDS(postprandial distress syndrome) Patients admitted to outpatient department with symptoms meeting ROME III criteria

SUMMARY:
There has been recent interest into the potential role of mucosal barrier defects in the pathophysiology of functional gastrointestinal disorders (FGIDs). There has been evidence of increased intestinal permeability in patients of IBS,and abnormal tissue resistance in NERD. Although the mucosa of Functional dyspepsia (FD) patients is endoscopically and histologically "normal," it contains ultrastructural changes, activated immune cells, along with evidence of an increased release of mediators leading to gastric dysfunction. There is now consistent evidence indicating that mucosal barrier defects allow the passage of an increased load of bacteria, antigens and toxins which, in turn evoke activation of mucosal immune responses involved in the FD symptom.

DETAILED DESCRIPTION:
Confocal laser endomicrosopy is a newly developed device which allows in vivo and real time observation of gastrointestinal mucosa.In our pilot study we found that the contrast agent fluorescein sodium shew differences of leakage into intercellular spaces and crypt lumen among different patients of FD.

This study is aimed to determine if there is microscopic changes detectable in the gastric mucosal epithelium through confocal endomicroscopy of FD patients, and to evaluate the relationship among minimal changes(transmission electron microscopy and Confocal laser endomicrosopy ), FD symptoms(symptom index form) , neuropeptides and immune responses(immunohistochemistry).

ELIGIBILITY:
Inclusion Criteria:

* patients meeting IBS diagnosis criteria and indications for endoscopy investigation.
* Asymptomatic individuals for health surveillance or patients for follow up after polypectomy.

Exclusion Criteria:

* Esophageal, gastric or duodenal cancer or other malignancy
* History of esophagus, stomach, or duodenum surgery
* Conditions that preclude safe biopsies (coagulopathy, haemophilia, esophageal varices,and patients on warfarin and antiplatelets)
* A history of bronchial asthma, or known allergy to fluorescein
* Pregnant or breast-feeding (for females)
* Below 18 or above 75 years of age
* Severe co-morbidities
* Unable or unwilling to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with indications for upper-endoscopy in Qilu Hospital outpatient and inpatient department are the study population of this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Specific microscopic changes in the gastric mucosa as seen under the confocal endomicroscope | Within the 30 minutes after injection of fluorescein

SECONDARY OUTCOMES:
the relationship among minimal changes, FD symptoms , neuropeptides and immune responses. | after the immunohistochemistry of biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China